CLINICAL TRIAL: NCT02969161
Title: Safe Generations Plus: Mother Infant Retention Across the Option B-plus Cascade
Brief Title: Safe Generations Plus: Swaziland PMTCT LTF Study
Acronym: SG+
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Ministry of Health, Swaziland (Other Government)
Responsible Party: Principal Investigator, William Reidy, Associate Research Scientist, ICAP, Columbia University
Other Study IDs: AAAP5700
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: PMTCT (Prevention of Mother-to-Child Transmission); HIV (Human Immunodeficiency Virus); Loss to follow-up (LTF); Option B+ (B+); ART (antiretroviral therapy)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to understand how to improve retention in care and treatment services to HIV positive pregnant women and their babies in Swaziland. The investigators will evaluate outcomes of patients who are lost-to-follow-up (LTF) under a new approach for prevention of mother-to-child (PMTCT) called Option B+, where all HIV positive pregnant women initiate lifelong antiretroviral therapy (ART) regardless of their disease stage. The goal is to understand the outcomes of patients who are LTF from care, and the reasons for disengagement from care in the context of PMTCT in order to inform efforts to improve retention in care among patients under Option B+.

DETAILED DESCRIPTION:
The study will be conducted among approximately 1,600 women and their infants who received Option B+ PMTCT services at ten facilities in Swaziland. These facilities were included in another study on Option B+ called Safe Generations in which routinely collected patient-level data was abstracted from medical registers. This study has three parts: the first is a review of alternative patient medical records among women and their infants who were documented as LTF in the Safe Generations study. The second component consists of tracing women who are LTF on the phone or in the community to administer a questionnaire. Lastly, an in-depth interview will be conducted among a sub-group of women to explore patterns of care.

ELIGIBILITY:
Inclusion Criteria:

* Mothers and their infants who were enrolled in PMTCT at Safe Generations study sites after the sites transitioned to Option B+.
* Determined to be LTF per the Safe Generations study protocol (i.e., have not attended a clinic visit in the 90 days prior to their 6-month postpartum appointment and are not known to be dead or transferred out, according to clinical visit data abstracted to the Safe Generations study database).

Exclusion Criteria:

* Mothers that are not a PMTCT client.

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV-infected pregnant mothers enrolled in PMTCT care under Option B+ as part of the Safe Generations study between September 16, 2013 and August 31, 2014
Sampling Method: Non-Probability Sample
Enrollment: 616 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are retained in care | Up to 24 months
  Confirmation of retained status among all Option B+ mothers and their infants who are identified as LTF per the Safe Generations study through review of facility-based records - to determine maternal reasons for leaving care.

SECONDARY OUTCOMES:
Proportion of patients who have died | Up to 24 months
  Confirmation patients being retained in care among all Option B+ mothers and their infants who are identified as LTF per the Safe Generations study through review of facility-based records - to capture events such as fetal loss and maternal/infant deaths that are not well documented.
Proportion of patients who are in care at another facility | Up to 24 months
  Mothers and/or infants who are LTF will be traced via telephone by facility-based healthcare workers or via questionnaire/interview conducted in the community - to determine if they have transferred care to another facility (via a self-transfer of care) and therefore remain engaged in care.
Proportion of patients who have disengaged from care entirely | Up to 24 months
  Confirmation of LTF status among all Option B+ mothers and their infants who are identified as LTF per the Safe Generations study through review of facility-based records - to capture events such as fetal loss and maternal/infant deaths that are not well documented.

CONTACTS AND LOCATIONS:
Overall Officials: William Reidy, PhD, Principal Investigator — ICAP at Columbia University; Elaine Abrams, PhD, Study Director — ICAP at Columbia University; Averie Gachuhi, MSc, Study Director — ICAP at Columbia University; Harriet Nuwagaba-Biribonwoha, MBChB, PhD, Study Director — ICAP at Columbia University
Locations (10):
- Eswatini (10):
  - Family Life Association Swaziland (FLAS) Manzini, Swaziland
  - King Sobhuza II Hospital, Swaziland
  - Luyengo Clinic, Swaziland
  - Mankayane PHU, Swaziland
  - Mbikwakhe Clinic, Swaziland
  - Médecins sans Frontières (MSF) Matsapha, Swaziland
  - Raleigh Fitkin Memorial Hospital, Swaziland
  - Siphofaneni Clinc, Swaziland
  - Siteki PHU, Swaziland
  - Lamvelase, Zombodze

IPD SHARING:
Plan to Share IPD: No